CLINICAL TRIAL: NCT03326375
Title: Comparison of Stereotactic Body Radiation Therapy (SBRT)and Repeat Transarterial Chemoembolization (TACE) for Hepatocellular Carcinoma (HCC) as a Local Salvage Treatment After Incomplete TACE : A Prospective Randomized Trial
Brief Title: Comparison of SBRTand Repeat TACE for HCC
Acronym: STH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Gangneung Asan Hospital (Other)
Collaborators: Soonchunhyang University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GNH_RT-001
Record Dates: First submitted 2017-04-24; First posted 2017-10-31 (Actual); Last update posted 2017-10-31 (Actual); Status verified 2017-10

CONDITIONS: HepatoCellular Carcinoma
Keywords: TACE; SBRT
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiosurgery

STUDY DESIGN:
Masking Description: open labled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SBRT (Stereotatic body radiotherapy) (Experimental): Treatment of SBRT in HCC patients who have incomplete response after first TACE
  Interventions: Radiation: SBRT
- TACE (Transarterial chemoembolization) (No Intervention): Treatment of repeated TACE in HCC patients who have incomplete response after first TACE

INTERVENTIONS:
Radiation: SBRT — Maximum dose : 60Gray (Gy) Fraction : 2 to 5
  Other Names: Stereotactic Body Radiation Therapy
  Arms: SBRT (Stereotatic body radiotherapy)

SUMMARY:
Comparison of Stereotactic Body Radiation Therapy (SBRT) and repeated transarterial chemoembolization (TACE) for Hepatocellular Carcinoma (HCC)as a Local Salvage Treatment after first incomplete TACE

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of SBRT after first incomplete TACE.

In HCC patients with incomplete TACE response, repeated TACE did not showed good response. In this case, SBRT could have better results than TACE.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Eastern cooperative oncology group(ECOG) score 0 to 2
* Primary HCC
* HCC (single nodule ≤ 7 cm or max 3 nodules ≤ 3 cm)
* Child-Turgottei-Pugh A or B
* Unresectable lesion or medically contraindicated surgery or a case in which surgery was declined.
* No evidence of radiologically definable major vascular invasion or extrahepatic disease
* Previously incomplete TACE with radiologically defined residual disease after first TACE
* Informed consent

Exclusion Criteria:

* Prior TACE to the target lesion
* Contraindication to receiving radiotherapy or TACE
* Decompensated liver cirrhosis
* Extrahepatic mets
* Pregnancy
* Patients with other cancers

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Local tumor control (efficacy fo SBRT) | 1 year
  To evaluate the effect of SBRT. Local tumor control is defined as the disappearance of any intraarterial enhancement in all target lesions.
  Local tumor control will be measured on triphasic Computerized Tomography (CT) or Magnetic Resonance Imaging (MRI). Patient will be asked to visit their study doctor for follow-up exams and imaging (CT or MRI) every 3 months.

SECONDARY OUTCOMES:
progression free-survival | 2 year
  survival from SBRT to recurrence
overall survival | 2 year
  survival from SBRT to death
Radiation induced liver disease (RILD) | 1 year
  Liver toxicities were evaluated using Common Terminology Criteria of Adverse Events (CTCAE).
  RILD was defined as elevated liver transaminases more than five times the upper normal limit or a worsening of Child-Pugh (CP) score by 2 within 3 months after SBRT.

CONTACTS AND LOCATIONS:
Overall Officials: Gab Jin Cheon, M.D, Ph. D, Study Director — University of Ulsan College of Medicine, Gangneung Asan Hospital
Locations (1):
- Gangneung Asan Hospital, Wŏnju, Gangwondo, South Korea

IPD SHARING:
Plan to Share IPD: No